CLINICAL TRIAL: NCT04519749
Title: An Open-label, Phase 1/2 Trial of Gene Therapy 4D-310 in Adults With Fabry Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4D-310-C001
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Fabry Disease
Keywords: Lysosomal Storage Diseases; Nervous System Brain Diseases; Metabolic; Inborn Brain Diseases; Metabolic Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cerebral Small Vessel Diseases; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Genetic Diseases; X-Linked; Inborn; Metabolic Diseases; Lipid Metabolism Disorders; Sphingolipidoses; Metabolism; Inborn Errors; Lipidoses; Lipid Metabolism
MeSH Terms: conditions — Fabry Disease; Lysosomal Storage Diseases; Brain Diseases, Metabolic; Central Nervous System Diseases; Nervous System Diseases; Cerebral Small Vessel Diseases; Cerebrovascular Disorders; Vascular Diseases; Cardiovascular Diseases; Genetic Diseases, Inborn; Metabolic Diseases; Lipid Metabolism Disorders; Sphingolipidoses; Lipidoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 4D-310 Dose Level 1 - AAV Neutralizing Antibody (NAb) Group A (Experimental): Single IV administration of 4D-310 Dose Level 1 - AAV NAb Titer Group A patients
  Interventions: Biological: 4D-310
- 4D-310 Dose Level 1 - AAV NAb Titer Group B (Experimental): Single IV administration of 4D-310 Dose Level 1 - AAV NAb titer Group B patients
  Interventions: Biological: 4D-310
- 4D-310 Dose Level 2 - AAV NAb Titer Group A and/or B (Experimental): Single IV administration of 4D-310 at Dose Level 2 in AAV NAb titer Group A and/or B patients
  Interventions: Biological: 4D-310
- 4D-310 Dose Expansion (Experimental): Dose expansion cohort of single IV administration of 4D-310 at the selected dose and selected AAV Nab titer group(s) patients
  Interventions: Biological: 4D-310

INTERVENTIONS:
Biological: 4D-310 — 4D-310 is a novel adeno-associated virus (AAV) gene therapy comprised of two active components: the capsid (4D-C102) and the transgene cassette, which encodes a codon-optimized full length human GLA transgene driven by the CAG promoter. 4D-310 has been engineered so that it cannot replicate (replication incompetent).

SUMMARY:
This is a prospective multicenter, open-label, dose-escalation trial to assess the safety, tolerability, and pharmacodynamics of 4D-310 following a single IV administration. The study population is comprised of adult males and females with Fabry Disease.

DETAILED DESCRIPTION:
This is a prospective multicenter, open-label, dose-escalation trial to assess the safety, tolerability, and pharmacodynamics of 4D-310 following a single IV administration. The study population is comprised of adult males and females with Fabry Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Pathogenic GLA mutation consistent with Fabry Disease
3. Confirmed diagnosis of classic or late-onset Fabry disease
4. Individuals on ERT must be on a stable dose for at least 6 months (and a minimum of 12 months total exposure) prior to study enrollment
5. Agree to use highly effective contraception

Exclusion Criteria:

1. Presence of high titer neutralizing antibody to 4D-310 capsid, or presence of high antibody titer to AGA
2. eGFR <45 mL/min/1.73 m2
3. Undergone kidney transplantation or currently on hemodialysis or peritoneal dialysis
4. HIV, active or chronic hepatitis B or C,
5. Evidence of liver disease, severe pulmonary disease or diabetes with poor glycemic control
6. History of stroke or transient ischemic attack within the last 12 months, or other significant thromboembolic disease history (e.g. pulmonary embolism)
7. Contraindication to systemic corticosteroid therapy or immunosuppressive therapy
8. Chronic steroid use, defined as ≥ 3 months of oral corticosteroid use within the last 12 months.
9. Moderately severe to severe cardiovascular disease or uncontrolled hypertension
10. Left ventricular ejection fraction of <45% on echocardiogram (ECHO)
11. Currently receiving investigational drug, device or therapy or having ever received gene therapy
12. History of infusion related response to ERT or any adverse reaction leading to ERT discontinuation
13. History of cancer within 2 years (exceptions include non-melanoma skin cancer, localized prostate cancer treated with curative intent)
14. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 1 year
  Safety and tolerability of 4D-310 following a single IV dose, as assessed by incidence and severity of adverse events, serious adverse events and dose limiting toxicities, including clinically significant changes from baseline to scheduled time points in safety parameters

SECONDARY OUTCOMES:
Change from baseline in serum AGA activity | 1 year
  Change from baseline in serum AGA activity
Change from baseline serum globotriaosylsphingosine (lysoGb3) | 1 year
  Change from baseline serum globotriaosylsphingosine (lysoGb3)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Cohen, MD, Study Director — 4D Molecular Therapeutics
Locations (4):
- United States (4):
  - University of California at San Diego, La Jolla, California
  - Emory University, Atlanta, Georgia
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Lysosomal & Rare Disorders Research & Treatment Center, Inc, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No